CLINICAL TRIAL: NCT04774432
Title: Effect of Granulocyte Macrophage Colony Stimulating Factor (GM-CSF) on Human in Vitro Oocyte Maturation (CAPA-IVM System) Success Rates in PCOS
Brief Title: Effect of GM-CSF on CAPA-IVM System Success Rates in PCOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01/21/DD-BVMD
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: IVF; PCOS; IVM
Keywords: GM-CSF; CAPA-IVM
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GM-CSF group (Active Comparator): Patients will be randomly allocated to intervention group with GM-CSF added to CAPA and maturation medium.
  Following the 24h CAPA period, the evaluation of maturation (MII, GVBD, GV) will be done after 30 hrs IVM step.
  Mature eggs are fertilized using Intracytoplasmic sperm injection (ICSI). Fertilized oocytes will be placed in a time-lapse incubator (ASTEC) and their development until the Day 5/6 (blastocyst formation) will be followed.
  Interventions: Other: GM-CSF group
- Control group (Active Comparator): Patients will be randomly allocated to control group without the addition of GM-CSF to CAPA and maturation medium.
  Following the 24h CAPA period, the evaluation of maturation (MII, GVBD, GV) will be done after 30 hrs IVM step.
  Mature eggs are fertilized using Intracytoplasmic sperm injection (ICSI). Fertilized oocytes will be placed in a time-lapse incubator (ASTEC) and their development until the Day 5/6 (blastocyst formation) will be followed.
  Interventions: Other: Control group

INTERVENTIONS:
Other: GM-CSF group — GM-CSF added to CAPA and maturation medium
  Arms: GM-CSF group
Other: Control group — GM-CSF will not be added to CAPA and maturation medium
  Arms: Control group

SUMMARY:
In-vitro maturation (IVM) of human oocytes obtained from minimally stimulated or unstimulated ovaries offers a more "patient friendly" treatment option than the conventional Assisted Reproductive Technology (ART) treatment with controlled ovarian hyperstimulation (COH). However, maturation rate and the total blastocyst yield in oocytes undergoing in vitro maturation are still limited.

This pilot study aims to evaluate the addition of an important growth factor known as Granulocyte macrophage colony stimulating factor (GM-CSF). The investigators hypothesize that the addition of GM-CSF to human IVM culture media will increase pregnancy rates to comparable levels to that of IVF, making it a viable clinical option for couples undergoing assisted reproductive treatment.

DETAILED DESCRIPTION:
In-vitro maturation (IVM) of human oocytes obtained from minimally stimulated or unstimulated ovaries offers a more "patient friendly" treatment option than the conventional Assisted Reproductive Technology (ART) treatment with controlled ovarian hyperstimulation (COH).

Typically, IVM will be offered to women with polycystic ovaries (PCO/PCOS), or to patients with an excellent ovarian reserve, i.e. a high antral follicle count. IVM treatment is characterized by minimal administration of FSH or HMG and NO HCG ovulation trigger.

The IVM approach is less disruptive to patients' daily life through the reduced need for hormonal and ultrasound monitoring, avoids a range of minor and major complications, such as ovarian hyperstimulation syndrome, and aims to reduce the total cost of infertility treatment for the patient and for the health care budget.

Human oocytes retrieved from small antral follicles are able to resume meiosis by undergoing germinal vesicle breakdown and extrusion of the first polar body, if they have reached meiotic competence. These oocytes can be fertilized although only a proportion (less than 50%) of them can develop further into viable embryos. It has been hypothesized that failure of embryonic development may, at least in part, be due to an immature oocyte cytoplasm.

The investigators have developed a novel human in vitro maturation (IVM) culture system (named CAPACITATION-IVM , hereafter named "CAPA") using 1°) natural compounds known to influence cGMP and cAMP levels within the cumulus-oocyte-complex and 2°) compounds that are crucial for the oocyte-cumulus cross-talk. Keeping cyclic AMP high after retrieval in the GV oocyte prevents occurrence of nuclear maturation, enabling increased communication between the oocyte and the cumulus cells. This allows for the improvement in the synchronization of nuclear and cytoplasmic maturation processes in the oocyte, to the benefit of embryo quality.

The clinical outcomes of using CAPA-IVM in PCOS instead of fully stimulated GnRH-antagonist HP-HMG stimulated IVF-ICSI treatments showed equivalent live-birth rates after a first embryo transfer cycle done in artificial endometrial preparation in the two arms. Nevertheless, the CAPA-IVM cumulative live birth at 12 months was 44%, while in IVF it was 62,6. (Vuong et al., 2020). Hence the attrition rate of embryos in CAPA-IVM is larger than in conventional ART. In order to correct for this difference in good embryo number there is a need to refine the culture conditions.

This pilot study aims to evaluate the addition of an important growth factor known as Granulocyte macrophage colony stimulating factor (GM-CSF). In a recent breakthrough it has been shown that adding GM-CSF to IVM media can improve preimplantation embryo development in pigs, cattle and mice (unpublished results from Prof Mark Nottle, Adelaide University, Australia). Moreover, in mice, these improvements lead to an increased in implantation rate (+62%) and tended to increase birth rate (+25%) following the transfer of vitrified/warmed blastocysts compared with standard IVM. Based on these findings, this pilot study aims to determine the beneficial effect of using GM-CSF during the biphasic CAPA-IVM. The investigators hypothesize that the addition of GM-CSF to human IVM culture media will increase pregnancy rates to comparable levels to that of IVF, making it a viable clinical option for couples undergoing assisted reproductive treatment.

GM-CSF (Leukine in EmbryoGene medium, Medicult) has previously been used as an additive in embryo culture in order to increase the implantation rate of exposed embryos. This study in more than 1000 patients showed no advantage of adding GMCSF routinely. However in a subset of patients, those with poor implantation, the addition of this factor improved clinical results (Ziebe et al., 2013). In this study no safety issues were mentioned by exposing human oocytes during fertilization and early embryo formation.

In the intended study there will be only exposure of GM-CSF during the oocyte maturation steps, and the embryos will never be in direct contact with the investigational compound.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as PCOS using Rotterdam criteria (AFC=25 or the ovarian volume >10ml)
* Agree to participate in the study

Exclusion Criteria:

* No major uterine or ovarian abnormalities
* Endometriosis grade 2 or upper
* Severe OAT (concentration <1 million/ml, motility <10%), surgical sperm

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-03-02 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Blastulation rate | At least seven days after oocyte pick up
  Percentage of blastocyst by 2 types of IVM culture with or without GM-CSF

SECONDARY OUTCOMES:
Embryology data (maturation rate, fertilization rate, grade 1 and grade 2 blastocyst rate) | Maturation rate: 2 days after OPU, Fertilization rate: 3 days after OPU, grade 1 and 2 blastocyst: at least 7 days after OPU
  Maturation rate: percentage of mature oocyte over oocytes pick-up by 2 types of IVM culture Fertilization rate: percentage of 2PN over oocytes injected by 2 types of IVM culture Grade 1 and 2 blastocyst rate: percentage of grade 1 and 2 blastocyst over total number of blastocysts by 2 types of IVM culture
Ongoing Pregnancy Rate after the first transfer of the started treatment cycle. | At 12 weeks' gestation
  Ongoing pregnancy is defined as pregnancy with detectable heart rate at 12 weeks' gestation or beyond, after the completion of the first transfer.
Cumulative ongoing pregnancy rate at 6 months after randomization | At 12 weeks' gestation at 6 months after randomization. After 6 months, most patients doing IVM have finished all their frozen embryos; therefore, we consider this time point for analyzing the cumulative ongoing pregnancy rate.
  Ongoing pregnancy is defined as pregnancy with detectable heart rate at 12 weeks' gestation or beyond, after transfer of all embryos from the started treatment cycle.
Adverse events (OHSS rate, miscarriage rate, ectopic rate) | OHSS rate: at 03 days after oocytes pick-up and 14 days after embryo transfer, Miscarriage rate: Before 22 weeks of gestational age, ectopic rate: At 5-7 weeks of gestation
  OHSS rate: Routine assessments for OHSS were performed on day 3 post oocyte retrieval in both groups. At other times, OHSS was evaluated if symptoms were reported by the patient. OHSS was classified using the flow diagram developed by Humaidan and colleagues for use in clinical trial settings Miscarriage defined as spontaneous loss of a clinical pregnancy before week 22 of gestational age, in which the embryo(s) or fetus(es) is/are nonviable and is/are not spontaneously absorbed or expelled from the uterus.
  Ectopic pregnancy defined as a pregnancy in which implantation takes place outside the uterine cavity
The relative expression ratio ( R ) of human cumulus cell genes | cumulus cells will be collected after at least 30 hours of maturation culture, storaged at -80oC until RNA purification
  Cumulus cells (CCc) will be collected, cDNA synthesis after mRNA purification, relative quantification PCR for detecting gene expression between CCs of GM-CSF group and CCs of control group.
Infant DNA methylation expression level | At the time of delivery
  Newborn's material (cord blood, buccal smears, placental tissue) will be collected for epigenetics analysis.
  Computational pipeline for genome-wide bisulfite sequencing data analysis. Reads from bisulfite sequencing are first aligned to the reference genome. The alignment data may be visualized in different tracks for comparison (control group vs GM-CSF group). After methylation calling, the bulk methylation level and genome-wide methylation level are calculated and plotted, and DMRs (differentially methylated regions) are determined. To perform an integrative analysis, DNA methylation data are coupled with gene expression, e.g., differentially genes (DEGs), to delineate the regulatory role of DNA methylation.

CONTACTS AND LOCATIONS:
Overall Officials: Tuong M Ho, MD, Principal Investigator — Hope Research Center
Locations (1):
- My Duc Hospital, Ho Chi Minh City, Vietnam

REFERENCES:
- [Background] Guzman L, Ortega-Hrepich C, Albuz FK, Verheyen G, Devroey P, Smitz J, De Vos M. Developmental capacity of in vitro-matured human oocytes retrieved from polycystic ovary syndrome ovaries containing no follicles larger than 6 mm. Fertil Steril. 2012 Aug;98(2):503-7.e1-2. doi: 10.1016/j.fertnstert.2012.01.114. Epub 2012 Feb 23. PMID 22365339
- [Background] Guzman L, Adriaenssens T, Ortega-Hrepich C, Albuz FK, Mateizel I, Devroey P, De Vos M, Smitz J. Human antral follicles <6 mm: a comparison between in vivo maturation and in vitro maturation in non-hCG primed cycles using cumulus cell gene expression. Mol Hum Reprod. 2013 Jan;19(1):7-16. doi: 10.1093/molehr/gas038. Epub 2012 Sep 6. PMID 22956770
- [Background] Heijnen EM, Eijkemans MJ, Hughes EG, Laven JS, Macklon NS, Fauser BC. A meta-analysis of outcomes of conventional IVF in women with polycystic ovary syndrome. Hum Reprod Update. 2006 Jan-Feb;12(1):13-21. doi: 10.1093/humupd/dmi036. Epub 2005 Aug 25. PMID 16123051
- [Background] Sanchez F, Lolicato F, Romero S, De Vos M, Van Ranst H, Verheyen G, Anckaert E, Smitz JEJ. An improved IVM method for cumulus-oocyte complexes from small follicles in polycystic ovary syndrome patients enhances oocyte competence and embryo yield. Hum Reprod. 2017 Oct 1;32(10):2056-2068. doi: 10.1093/humrep/dex262. PMID 28938744
- [Background] Ho VNA, Braam SC, Pham TD, Mol BW, Vuong LN. The effectiveness and safety of in vitro maturation of oocytes versus in vitro fertilization in women with a high antral follicle count. Hum Reprod. 2019 Jun 4;34(6):1055-1064. doi: 10.1093/humrep/dez060. PMID 31111879
- [Background] Ziebe S, Loft A, Povlsen BB, Erb K, Agerholm I, Aasted M, Gabrielsen A, Hnida C, Zobel DP, Munding B, Bendz SH, Robertson SA. A randomized clinical trial to evaluate the effect of granulocyte-macrophage colony-stimulating factor (GM-CSF) in embryo culture medium for in vitro fertilization. Fertil Steril. 2013 May;99(6):1600-9. doi: 10.1016/j.fertnstert.2012.12.043. Epub 2013 Feb 4. PMID 23380186